CLINICAL TRIAL: NCT05531071
Title: Clinical Observation of Acupuncture Combined With Biofeedback Electrical Stimulation in the Treatment of Female Stress Urinary Incontinence
Brief Title: Effect of Acupuncture Combined With Biofeedback Electrical Stimulation on SUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei General Hospital (Other)
Responsible Party: Principal Investigator, Caiqing Ji, head nurse, Hebei General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HebeiGH
Record Dates: First submitted 2022-08-31; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary incontinence; Acupuncture; Biofeedback electrical stimulation
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biofeedback electrical stimulation (Active Comparator): Use the PHENIX USB4 Pelvic Floor Rehabilitation Therapy Apparatus to enter the Stress Urinary Incontinence Treatment Module. The frequency of electrical stimulation was 50Hz, the pulse width was 250μs, and the current intensity increased from 0mA, generally not exceeding 50mA. For the 1st to 3rd treatments, intermittent bioelectrical stimulation mode was given.For the 4th to 10th treatments, the biofeedback mode with intermittent bioelectrical stimulation was given, and for the 11th to 15th treatments, the simple biofeedback mode was given. 3 times a week, 30 minutes each time, a total of 15 treatments. Instruct the patient to go home to perform pelvic floor muscle training, focusing on anal contractions. Each anal contraction takes 3-5s and relaxes for 5-10s. so repeatedly. 20 minutes each time, 3 times a day in the morning, noon and evening, 5 days a week, until the end of the treatment.
  Interventions: Device: Biofeedback electrical stimulation
- Acupuncture (Active Comparator): A single-use sterile needle of Changchun Aikang brand was selected, with a size of 0.30 mm × 40 mm. Ding points: Guanyuan point, Qihai point, Zhongji point, Zusanli point, Sanyinjiao point, Yinlingquan point. Routine disinfection of the patient's skin is performed, and Guanyuan, Qihai, and Zhongji points are punctured obliquely downward, and the needle is inserted 1-1.2 cun; evenly lift, insert and twist to get qi. At the same time, the moxa column was ignited and placed in the moxibustion box, and the moxibustion box was placed above the three points of Guanyuan, Qihai, and Zhongji in the patient's abdomen, and the moxibustion was performed until the skin was red and the deep tissue was heated. 1 time a day, every Monday to Friday, 30 minutes each time, 10 times as a course of treatment. The patients were instructed to go home for pelvic floor muscle training, and the method was the same as that of group Biofeedback electrical stimulation.
  Interventions: Procedure: Acupuncture
- Acupuncture combined with biofeedback electrical stimulation (Experimental): Biofeedback electrical stimulation therapy combined with acupuncture and moxibustion were given to the patients. After 10 sessions of acupuncture, continue the unfinished biofeedback electrical stimulation treatment. The patients were instructed to go home for pelvic floor muscle training, and the method was the same as that of group Biofeedback electrical stimulation.
  Interventions: Combination Product: Acupuncture combined with biofeedback electrical stimulation

INTERVENTIONS:
Device: Biofeedback electrical stimulation — treated with biofeedback electrical stimulation, 3 times a week for 30 minutes for 15 times.
  Arms: Biofeedback electrical stimulation
Procedure: Acupuncture — acupuncture treatment, including Guanyuan, Qihai, Zhongji, Zusanli, Sanyinjiao and Yinlingquan, once a day, Monday to Friday, 30 minutes each, a total of 10 times.
  Arms: Acupuncture
Combination Product: Acupuncture combined with biofeedback electrical stimulation — treated with acupuncture combined with biofeedback electrical stimulation.
  Arms: Acupuncture combined with biofeedback electrical stimulation

SUMMARY:
Objective: To investigate the clinical efficacy of acupuncture combined with biofeedback electrical stimulation on female stress urinary incontinence. Methods: 90 patients diagnosed in a hospital from January 2020 to January 2021 were randomly divided into three groups A, B and C, and group A was treated with biofeedback electrical stimulation, 3 times a week for 30 minutes for 15 times. Group B used acupuncture treatment, including Guanyuan, Qihai, Zhongji, Zusanli, Sanyinjiao and Yinlingquan, once a day, Monday to Friday, 30 minutes each, a total of 10 times. Group C was treated with acupuncture combined with biofeedback electrical stimulation. All three groups were combined with pelvic floor muscle training. After treatment, the changes in class I, II muscle fiber, ICI-Q-SF score, and urine leakage in the 1h pad test were compared.

ELIGIBILITY:
Inclusion Criteria:

* meet the diagnostic criteria of SUI
* Aged over 18 years old and have a history of sexual life
* No treatment related to SUI within three months
* Mental illness without cognitive dysfunction, able to cooperate with examination and treatment
* Voluntarily participate and sign the informed consent

Exclusion Criteria:

* combined with urge urinary incontinence, uterine prolapse, vaginal anterior and posterior wall prolapse
* pregnancy, postpartum lochia or abnormal vaginal bleeding
* Acute phase of inflammation (pelvic cavity, vagina, urinary system)
* There are metal substances such as pacemakers and metal stents in the body
* Denervation of pelvic floor muscles (no sensation, no contraction)
* coagulation dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle strength | Before treatment
  Use the French Sugiyama PHENIX USB2 pelvic floor rehabilitation therapy instrument to detect the muscle strength of pelvic floor type I muscle fibers and type II muscle fibers. Class I muscle strength: amplitude height ≥ 40%, duration 0-5s corresponds to 0-5 level muscle strength; Class II muscle strength: Amplitude height ≥ 60%, 0 to 5 times of duration corresponds to 0 to 5 levels of muscle strength.
Pelvic floor muscle strength | 4 weeks
  Use the French Sugiyama PHENIX USB2 pelvic floor rehabilitation therapy instrument to detect the muscle strength of pelvic floor type I muscle fibers and type II muscle fibers. Class I muscle strength: amplitude height ≥ 40%, duration 0-5s corresponds to 0-5 level muscle strength; Class II muscle strength: Amplitude height ≥ 60%, 0 to 5 times of duration corresponds to 0 to 5 levels of muscle strength.
1 hours urine pad test | Before treatment
  the patient empties the bladder before the test, and the urine pad is weighed and placed in the perineum. 0-15minutes, the patient drinks the mineral water prepared in advance; 16-45minutes, the patient walks as usual, going up and down the stairs; 46-60minutes, the patient runs on the spot for 1 minutes, sits up continuously, coughs forcefully 10 times, and bends over Take the action 5 times, and finally wash your hands with tap water for 1 minutes. After 1hours, the patient was instructed to take out the urine pad and weigh it, retain the urine and measure the urine volume. Urine leakage ≥ 2g is positive; according to the amount of urine leakage, the degree of urinary incontinence can be divided: 2g≤urine leakage <5g is mild, 5≤urine leakage <10g is moderate, 10g≤urine leakage <50g is severe, Urine leakage ≥ 50g is considered extremely severe.
1 hours urine pad test | 4 weeks
  the patient empties the bladder before the test, and the urine pad is weighed and placed in the perineum. 0-15minutes, the patient drinks the mineral water prepared in advance; 16-45minutes, the patient walks as usual, going up and down the stairs; 46-60minutes, the patient runs on the spot for 1 minutes, sits up continuously, coughs forcefully 10 times, and bends over Take the action 5 times, and finally wash your hands with tap water for 1 minutes. After 1hours, the patient was instructed to take out the urine pad and weigh it, retain the urine and measure the urine volume. Urine leakage ≥ 2g is positive; according to the amount of urine leakage, the degree of urinary incontinence can be divided: 2g≤urine leakage <5g is mild, 5≤urine leakage <10g is moderate, 10g≤urine leakage <50g is severe, Urine leakage ≥ 50g is considered extremely severe.
International Consultation on Incontinence Questionnaire short form | 4 weeks
  The patients reviewed their situation in the last 4 weeks, and scored three questions: the frequency of urine leakage, the amount of urine leakage, and the degree of impact on daily life. The minimum and maximum values were 0 and 21 respectively. The higher the total score, the more severe the symptoms of urinary incontinence, worse outcome. The greater the impact on life.

CONTACTS AND LOCATIONS:
Locations (1):
- Caiqing Ji, Shijiazhuang, Hebei, China